CLINICAL TRIAL: NCT04552275
Title: Circulating Biomarkers of Hypo-Attenuated Leaflet Thickening After Transcatheter Aortic Valve Replacement
Brief Title: The HALT Biomarker Study
Acronym: HALT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medtronic (Industry); Catholic Medical Center (Other); Minneapolis Heart Institute (Other)
Responsible Party: Principal Investigator, Sammy Elmariah, Director, Interventional Cardiology Research, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P001793
Record Dates: First submitted 2020-08-28; First posted 2020-09-17 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Aortic Stenosis; Hypo-attenuated Leaflet Thickening; Bioprosthetic Valve Degeneration
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HALT Cohort (Other): Patients who develop HALT
  Interventions: Diagnostic Test: Proteomics Analysis
- Control Group (Other): Patients who do not develop HALT
  Interventions: Diagnostic Test: Proteomics Analysis

INTERVENTIONS:
Diagnostic Test: Proteomics Analysis — Determine a panel of circulating proteins that discriminates between patients with and without Hypo-Attenuated Leaflet Thickening (HALT)

SUMMARY:
The purpose of the HALT Biomarkers study are to identify a panel of circulating proteins that discriminates between patients with and without Hypo-Attenuated Leaflet Thickening (HALT) and can be used to supplement the diagnosis of HALT; to characterize changes in circulating proteins after treatment of HALT with systemic anticoagulation; and to identify circulating proteins that predict the occurrence of HALT.

The study population will be adult patients undergoing transfemoral transcatheter aortic valve replacement (TAVR) for severe aortic stenosis (AS) or bioprosthetic valve degeneration. Enrollment will continue until 30 patients with HALT are identified for completion of phase 1. Based on a HALT incidence rate of 10%, we anticipate enrolling 300 patients.

Patients are enrolled prior to undergoing transfemoral TAVR. Blood samples, clinical data and echocardiograms will be collected at the following timepoints: baseline (pre-TAVR, T0), post-TAVR (pre-discharge, T1), 30-day follow-up (window 3-9 weeks, T2), and 6-month follow-up (T3). Cardiac 4D CT will be performed at the 30-day follow-up visit to screen for the occurrence of HALT.

Patients with HALT will be treated with systemic anticoagulation for 5-6 months, at which point a follow-up CT scan and blood sample will be obtained. Control subjects will also undergo a 6-month study visit with blood sample collection. The study will be conducted within two phases. Phase 1 will serve as a derivation / discovery study in which candidate protein biomarkers of HALT will be identified.

Once this is successfully completed, a second cohort will be enrolled within phase 2. Phase 2 will be performed under the auspices a future contract or amendment and will seek to cross-validate the initial study findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 65 years
2. Subject with severe native AS or severe bioprosthetic valve degeneration
3. Subject undergoing transfemoral TAVR using a Medtronic Evolut R, Evolut Pro or Evolut Pro+ transcatheter heart valve

Exclusion Criteria:

1. Chronic anticoagulation therapy
2. Contraindication to systemic oral anticoagulation therapy
3. Chronic kidney disease with EGFR<30 ml/min
4. Bleeding diathesis or known coagulopathy
5. Hypercoagulable state
6. Life-expectancy <12 months due to other medical conditions (e.g., malignancy, severe Alzheimer's disease, etc.)
7. The patient is currently participating in another investigational device or drug study that has not reached its primary objective/endpoint
8. Pregnant, lactating, or planning pregnancy within next 12 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2030-06-22 (Estimated); Study Completion 2035-06-22 (Estimated)

PRIMARY OUTCOMES:
Derivation of the panel of circulating proteins indicative of HALT | 6 months
  1. Establish the incidence of similar proteomic profiles and the rate to which the profile occurs in TAVR recipients with HALT via a high-throughput precision proteomics platform which utilizes the proximity extension assay (PEA). PEA merges a dual-recognition antibody-based immunoassay with quantitative real-time PCR that allows for the simultaneous quantification of 92 proteins. We will focus on the 5 highest yield panels for the current investigation: cardiovascular II, cardiovascular III, cardiometabolic, inflammation, and oncology II panels. These panels will allow for the assessment of 460 circulating proteins.
Establish the rate at which these characteristics indicative of future HALT | 6 months
  Using data analysis of baseline patient characteristics to establish the rate that they are indicative of future HALT in patients with aortic stenosis. The sampling frame assumes the sequencing of 460 proteins; a 5% False Discovery Rate; a 10% prognostic prevalence; a minimum fold change of 2; and a normalization ratio of 1.

SECONDARY OUTCOMES:
Cross-validation of the panel of circulating proteins indicative of HALT | 6 months
  3. Using 20 matched pairs of subjects with and without HALT, the derivation of the HALT indicative panel of circulating proteins gathered through PEA will be cross-validated using data analysis to establish the rate to which the panel is present in both cohorts. This rate will be used to determine if the proteomic profile of a patient can be used as a diagnostic test for the presence of HALT.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Catholic Medical Center, Manchester, New Hampshire

IPD SHARING:
Plan to Share IPD: No